CLINICAL TRIAL: NCT06380777
Title: Establishment and Application of a Digital Diagnosis and Treatment System for Sarcopenia
Brief Title: Establishment and Application of Digital Diagnosis and Treatment System for Sarcopenia
Status: Recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Yu Kang, MD, professor, Peking Union Medical College Hospital
Other Study IDs: DDT system for sarcopenia
Record Dates: First submitted 2024-04-06; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples Without DNA — blood and stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to establish a digital diagnosis and treatment system for sarcopenia, integrating research outcomes into a unified approach encompassing a digital vaccine (early warning screening model), digital drug (intervention model associated with pathogenesis), and digital rehabilitation (preventive system combining early warning and treatment). This aims to create a digital visual tertiary prevention network for sarcopenia.

Research aims:

Evaluate the effectiveness of the digital vaccine through a cross-sectional epidemiological survey.

Establish a specialized cohort for sarcopenia through a longitudinal investigation, implementing the digital drug and digital rehabilitation interventions.

Participants will:

Engage in screening and assessment based on inclusion and exclusion criteria.

Be monitored longitudinally, with tailored interventions for those with muscle atrophy and regular follow-ups for at-risk individuals.

Key outcomes will focus on sarcopenia indicators, serum biomarkers, and clinical endpoints such as fracture rates, weakness classification, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥45 years;
* meeting sarcopenia diagnostic criteria;
* consent to participate in this study

Exclusion Criteria:

* Age <45 years;
* patients in acute phase of chronic illness;
* infectious disease patients;
* people who lack of independent mobility;
* people who lack of communication or cognitive skills;
* people who refusal to participate in this study

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: outpatient patients, inpatients, elderly population in elderly care institutions, and community registered elderly patients in the north part of China
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Appendicular skeletal muscle mass index | Through study completion, an average of 6weeks
  Defined as muscle mass (Unit: kg/m2)

SECONDARY OUTCOMES:
Hand grip strength | Through study completion, an average of 6weeks
  Defined as muscle strength (Unit: kg)
Gait speed | Through study completion, an average of 6weeks
  Defined as physical performance (Unit: m/s)

OTHER OUTCOMES:
Concentration of insulin | Through study completion, an average of 6weeks
  Serum insulin levels
Concentration of adiponectin | Through study completion, an average of 6weeks
  Serum adiponectin levels
Concentration of leptin | Through study completion, an average of 6weeks
  Serum leptin levels
Concentration of insulin like growth factor -1(IGF-1) | Through study completion, an average of 6weeks
  Serum IGF-1 levels
Concentration of interleukin 18 (IL-18) | Through study completion, an average of 6weeks
  Serum IL-18 levels
Concentration of tumor necrosis factor - α (TNF-α) | Through study completion, an average of 6weeks
  Serum TNF-α levels
Concentration of TNF-like weak inducer of apoptosis (TWEAK) | Through study completion, an average of 6weeks
  Serum TWEAK levels
Concentration of fibroblast growth factor -19 (FGF-19) | Through study completion, an average of 6weeks
  Serum FGF-19 levels
Concentration of myostatin | Through study completion, an average of 6weeks
  Serum myostatin levels
Concentration of chemoattractant protein-1 (MCP-1) | Through study completion, an average of 6weeks
  Serum MCP-1 levels
Concentration of activin | Through study completion, an average of 6weeks
  Serum activin levels

CONTACTS AND LOCATIONS:
Overall Officials: Kang Yu, Study Director — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No